CLINICAL TRIAL: NCT04742530
Title: Effects of Extended Fasting Prior to Evening Exercise on Appetite, Energy Intake and Performance.
Brief Title: Fasted Evening Exercise: Performance and Compensatory Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham Trent University (Other)
Collaborators: Loughborough University (Other)
Responsible Party: Principal Investigator, Tommy Slater, Principle Investigator, Nottingham Trent University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TS_FastEvEx_2021
Record Dates: First submitted 2021-01-27; First posted 2021-02-08 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Obesity
Keywords: Fasted exercise; Energy intake; Energy balance; Appetite; Exercise performance
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The study design is a randomised, controlled, crossover design in which participants undertake three exercise conditions in a randomised order with at least a seven day period in between trials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fasted Evening Exercise (Experimental): Exercise will take place in the evening, following a 7 hour period of fasting.
  Interventions: Behavioral: Fasted Evening Exercise
- Fed Evening Exercise (Active Comparator): Exercise will take place in the evening, after having consumed a carbohydrate-containing meal 2 hours prior.
  Interventions: Behavioral: Fed Evening Exercise
- Fed Morning Exercise (Active Comparator): Exercise will take place in the morning, after having consumed a carbohydrate-containing meal 2 hours prior.
  Interventions: Behavioral: Fed Morning Exercise

INTERVENTIONS:
Behavioral: Fasted Evening Exercise — A 45 minute exercise session will take place on a stationary cycle ergometer at 18:30, after a 7-hour period of fasting. This will consist of 30 minutes of steady state cycling at 60% of VO2max, followed by an exercise test during which participants will complete as much work as they can within 15 minutes.
  Arms: Fasted Evening Exercise
Behavioral: Fed Evening Exercise — A 45 minute exercise session will take place on a stationary cycle ergometer at 18:30, after having consumed a carbohydrate-containing meal (20% estimated energy requirements) 2 hours prior. This will consist of 30 minutes of steady state cycling at 60% of VO2max, followed by an exercise test during which participants will complete as much work as they can within 15 minutes.
  Arms: Fed Evening Exercise
Behavioral: Fed Morning Exercise — A 45 minute exercise session will take place on a stationary cycle ergometer at 10:30, after having consumed a carbohydrate-containing meal (20% estimated energy requirements) 2 hours prior. This will consist of 30 minutes of steady state cycling at 60% of VO2max, followed by an exercise test during which participants will complete as much work as they can within 15 minutes.
  Arms: Fed Morning Exercise

SUMMARY:
This study will compare the appetite, energy intake, and exercise performance responses to a bout of exercise completed in the evening after an extended period of fasting with a similar bout of exercise completed in the evening and the morning, after consuming a carbohydrate-containing meal.

DETAILED DESCRIPTION:
Regular exercise is known to be a successful strategy for improving several facets of health and maintaining body weight. However, many people are not engaging in enough exercise, and some may not be achieving maximum benefits from the exercise that they already do. Performing exercise in the overnight fasted state has been shown to reduce energy intake over the course of a single day, without any compensatory reductions in free-living energy expenditure. Despite these promising findings, it is likely that not every member of the population is logistically able to perform exercise in the morning due to various work, family and social commitments, and exercise in the evening may be a logical alternative for these individuals. Whether the beneficial effects of overnight fasted exercise can be observed at an alternative time of the day (i.e. the evening) is unknown.

Therefore, the investigators are interested in examining the compensatory appetite and energy intake responses following a bout of evening exercise performed after an extended (7 hour) period of fasting. Exercise performance will also be assessed as a marker of voluntary energy expenditure, which if reduced, has the potential to compensate for the reduced energy balance induced by fasted exercise.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers.
* Have maintained a stable weight for 6 months (self-reported).
* No history of gastric, digestive, cardiovascular or renal disease (self-reported).
* Female specific: must be using a monophasic, low dose combined OCP (containing less than 50μg oestradiol and a synthetic progestin) OR females with regular menstrual cycles (self-reported).

Exclusion Criteria:

* Have an unusual eating pattern (i.e., extended fasting periods >8h other than overnight - self-reported).
* Severe food allergies, dislike or intolerance of study foods or drinks.
* Currently undergoing a lifestyle intervention (structured diet or exercise)
* Diagnosis of a condition or currently undergoing treatment therapy known to affect glucose or lipid metabolism (e.g., type-2 diabetes, taking statins), or contraindications to exercise.
* Use of medication or supplements that may affect hormone concentrations.
* Excessive alcohol consumption (>14 units/week).
* Intensive training schedule (>10 hours/week).
* Having received a positive COVID-19 test in the 6-month period prior to participation.
* Female specific: currently pregnant or breastfeeding, the use of any hormonal contraception, and the self-reporting of short (<24 d), long (>35 d), or irregular menstrual cycles.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Voluntary energy intake (Kilocalories) at a laboratory-based test meal | 15 minutes following the end of the exercise session.
  A laboratory-based meal consisting of pasta, tomato sauce and olive oil will be provided to participants in excess of expected consumption. Participants will be permitted 20 minutes to eat as much or as little as they desire, until 'comfortably full and satisfied'.
Exercise Performance (Voluntary Energy Expenditure) | Within the 15-minute performance test component of the exercise session.
  Maximum energy expenditure (Kilojoules) that can be completed within 15 minutes on a stationary bicycle ergometer. The participant will be able to alter their power output by selecting up or down on the ergometer control unit as they please.

SECONDARY OUTCOMES:
Visual Analogue Scale for Subjective Ratings of Appetite | Baseline, 2 hours, 3 hours, 3.5 hours, 5 hours, 7 hours, 8 hours, 10 hours, 11 hours, 12 hours, 14 hours, and 24 hours.
  Time-course of subjective ratings of hunger between breakfast provision and one hour after consuming lunch, measured using an appetite visual analogue scale. The scale is divided into subscales of different appetite perceptions including: hunger, fullness, desire to eat and prospective food consumption. Each subscale is rated on a 100mm scale (i.e. from 0 - 100), with a rating of 100 fully supporting the perception and a rating of 0 fully opposing the perception.
Substrate Utilisation During Steady State Exercise. | Within the 30-minute steady-state component of the exercise session.
  Measurements of VO2 and VCO2 during a 30 minute steady state bout of cycling which precedes the 15-minute performance test.
Rating of Perceived Exertion (RPE). | Within the 45-minute exercise session.
  RPE will be measured at 5-minute intervals throughout the 45-minute exercise period (30 min steady state; 15 min performance test) on a 6-20 RPE scale. The participant will point to the value that corresponds to their current perceived exertion (6 being no exertion at all; 20 being maximal exertion).
Enjoyment of the Exercise Bout | Immediately following the end of the exercise session.
  A shortened version of The Physical Activity Enjoyment Scale (PACES) will be completed to gauge enjoyment of the exercise sessions. A scale from 1-7 will be used for eight feelings. The participant will circle the value that corresponds to which (6 being no exertion at all; 20 being maximal exertion).
  The scale is divided into bipolar subscales of different feelings including: enjoyment, liking, pleasure, fun, pleasantness, interest, engagement and task absorption . Each subscale is rated on a 1-7 bipolar scale (i.e. from 1 - 7), with a rating of 1 fully supporting the feeling on the left-hand side of the subscale, and a rating of 7 fully supporting the feeling on the right-hand side of the subscale. For three subscales, a positive feeling is placed at 7, and for four subscales, a negative feeling is placed at 7 (reverse scored).
Pre-exercise Subjective Feelings | Immediately before the exercise session.
  A single questionnaire to assess pre-exercise subjective feelings will be measured using a visual analogue scale. The scale is divided into subscales of different feelings including: motivation, readiness, tiredness, nausea, and energetic. Each subscale is rated on a 100mm scale (i.e. from 0 - 100), with a rating of 100 fully supporting the perception and a rating of 0 fully opposing the perception.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Loughborough University, Loughborough
  - Nottingham Trent University, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Edinburgh RM, Hengist A, Smith HA, Travers RL, Betts JA, Thompson D, Walhin JP, Wallis GA, Hamilton DL, Stevenson EJ, Tipton KD, Gonzalez JT. Skipping Breakfast Before Exercise Creates a More Negative 24-hour Energy Balance: A Randomized Controlled Trial in Healthy Physically Active Young Men. J Nutr. 2019 Aug 1;149(8):1326-1334. doi: 10.1093/jn/nxz018. PMID 31321428
- [Background] Bachman JL, Deitrick RW, Hillman AR. Exercising in the Fasted State Reduced 24-Hour Energy Intake in Active Male Adults. J Nutr Metab. 2016;2016:1984198. doi: 10.1155/2016/1984198. Epub 2016 Sep 21. PMID 27738523
- [Background] Clayton DJ, Barutcu A, Machin C, Stensel DJ, James LJ. Effect of Breakfast Omission on Energy Intake and Evening Exercise Performance. Med Sci Sports Exerc. 2015 Dec;47(12):2645-52. doi: 10.1249/MSS.0000000000000702. PMID 25970668
- [Background] McIver VJ, Mattin LR, Evans GH, Yau AMW. Diurnal influences of fasted and non-fasted brisk walking on gastric emptying rate, metabolic responses, and appetite in healthy males. Appetite. 2019 Dec 1;143:104411. doi: 10.1016/j.appet.2019.104411. Epub 2019 Aug 21. PMID 31445052
- [Background] James LJ, Moss J, Henry J, Papadopoulou C, Mears SA. Hypohydration impairs endurance performance: a blinded study. Physiol Rep. 2017 Jun;5(12):e13315. doi: 10.14814/phy2.13315. PMID 28637708
- [Background] Metcalfe RS, Thomas M, Lamb C, Chowdhury EA. Omission of a carbohydrate-rich breakfast impairs evening endurance exercise performance despite complete dietary compensation at lunch. Eur J Sport Sci. 2021 Jul;21(7):1013-1021. doi: 10.1080/17461391.2020.1797890. Epub 2020 Aug 27. PMID 32674691
- [Background] Maffucci DM, McMurray RG. Towards optimizing the timing of the pre-exercise meal. Int J Sport Nutr Exerc Metab. 2000 Jun;10(2):103-13. doi: 10.1123/ijsnem.10.2.103. PMID 10861332
- [Background] Wallis GA, Gonzalez JT. Is exercise best served on an empty stomach? Proc Nutr Soc. 2019 Feb;78(1):110-117. doi: 10.1017/S0029665118002574. Epub 2018 Oct 18. PMID 30334499
- [Background] Kendzierski, D., & DeCarlo, K. J. (1991). Physical Activity Enjoyment Scale: Two Validation Studies. Journal of Sport and Exercise Psychology, 13(1), 50-64. doi:10.1123/jsep.13.1.50.
- [Background] Raedeke, T. D. (2007). The Relationship Between Enjoyment and Affective Responses to Exercise. Journal of Applied Sport Psychology, 19(1), 105-115. doi:10.1080/10413200601113638
- [Derived] Mode WJA, Slater T, Pinkney MG, Hough J, James RM, Varley I, James LJ, Clayton DJ. Effects of Morning Vs. Evening exercise on appetite, energy intake, performance and metabolism, in lean males and females. Appetite. 2023 Mar 1;182:106422. doi: 10.1016/j.appet.2022.106422. Epub 2022 Dec 17. PMID 36539157